CLINICAL TRIAL: NCT05192200
Title: AN OPEN LABEL, LONG-TERM EXTENSION STUDY TO INVESTIGATE THE SAFETY OF PF-06823859 ADMINISTERED TO ADULT PARTICIPANTS ≥18 AND ≤80 WITH ACTIVE DERMATOMYOSITIS.
Brief Title: An Extension Study for Participants Who Have Completed the Treatment Period of a Qualifying Parent Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C0251008; 2021-004787-10 (EudraCT Number)
Record Dates: First submitted 2021-12-01; First posted 2022-01-14 (Actual); Results first posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Dermatomyositis
MeSH Terms: conditions — Dermatomyositis

STUDY DESIGN:
Intervention Model Description: Eligible participants will have completed the treatment period of a qualifying Dermatomyositis parent study. All participants will receive active study drug.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Anti-Beta Interferon drug (PF-06823859) (Experimental): IV infusion
  Interventions: Drug: Anti-Beta Interferon (PF-06823859)

INTERVENTIONS:
Drug: Anti-Beta Interferon (PF-06823859) — IV infusion

SUMMARY:
The purpose of this research study is to evaluate the long-term safety, and tolerability of PF-06823859 study drug in adult participants with Dermatomyositis (DM) from a qualifying study.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged ≥18 and ≤80 with moderate to severe dermatomyositis (DM), that have completed the treatment period of a qualifying study.
* Capable of giving signed informed consent.
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.

Exclusion Criteria:

* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study
* Participants who met discontinuation criteria at any point during the participating qualifying studies.
* Participants with an ongoing safety event in the qualifying studies which, in the opinion of the investigator or sponsor, is an ongoing safety concern OR the participant has met safety monitoring criteria in the qualifying study that has not resolved.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (24):
- United States (20):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Alabama at Birmingham, Department of Dermatology, Birmingham, Alabama
  - Mayo Clinic, Scottsdale, Arizona
  - Attune Health Research Inc., Beverly Hills, California
  - Mayo Clinic in Florida, Jacksonville, Florida
  - KU Clinical Research Center - Clinical and Translational Science Unit (CTSU), Fairway, Kansas
  - KU Clinical and Translational Science Unit (CTSU) Rainbow, Kansas City, Kansas
  - University of Kansas Medical Center, Kansas City, Kansas
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital - CTH, Boston, Massachusetts
  - Center for Outpatient Health, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - NYU Grossman School of Medicine, The Ronald O. Perelman Department of Dermatology, New York, New York
  - NYU Langone Health Clinical Research Center, New York, New York
  - NYU Langone Radiology - Ambulatory Care Center East 41st Street, New York, New York
  - Mount Sinai Doctors Dermatology, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Center for Human Phenomic Science, Philadelphia, Pennsylvania
  - University of Pennsylvania, Perelman Center for Advanced Medicine (PCAM), Philadelphia, Pennsylvania
- Debreceni Egyetem Klinikai Kozpont, Debrecen, Hungary
- Poland (2):
  - Nova Reuma Społka Partnerska, Bialystok, Podlaskie Voivodeship
  - Centrum Medyczne Plejady, Krakow
- Hospital Universitario 12 de Octubre, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C0251008

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants with moderate to severe dermatomyositis (DM) who completed the treatment period of qualifying study C0251002 [NCT03181893] and had agreement from their study doctor to continue active treatment were enrolled in this study. A total of 24 participants (9 participants from the skin predominant cohort [Amended stage 2] and 15 participants from the muscle predominant cohort [Stage 3]) of the study C0251002 were enrolled in this open label, long-term extension (OLE) study.
Pre-assignment Details: As planned, in participant flow discontinuations were reported by treatment.
Groups:
- PF-06823859 600mg: All Participants: Participants with DM received PF-06823859 600 milligrams (mg) intravenously (IV) once every 4 weeks. The treatment duration was up to 48 weeks (treatment period was up through and including Week 52). There was a follow-up period of 16 weeks post treatment period, however participants were assessed for safety from Day 1 of treatment up to end of study (Week 68).
Period: Treatment Period
Arm/Group | PF-06823859 600mg: All Participants
Started | 24
Safety Analysis Set (All participants enrolled who took at least 1 dose of study intervention, regardless of which stage the participant entered from.) | 24
Skin Analysis Set (Participants with skin predominant DM who were enrolled in Amended Stage 2 of the C0251002 [NCT03181893] study and received at least 1 dose of study intervention.) | 9
Muscle Analysis Set (Participants with muscle predominant DM who were enrolled in Stage 3 of the C0251002 [NCT03181893] study and received at least 1 dose of study intervention.) | 15
Completed | 21
Not Completed | 3
Not completed — Other | 1
Not completed — Lack of Efficacy | 1
Not completed — Withdrawal by Subject | 1
Period: Follow-up
Arm/Group | PF-06823859 600mg: All Participants
Started | 22 (Participants who were followed-up)
Completed | 21
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants enrolled who took at least 1 dose of study intervention. This included all such participants regardless of which stage the participant entered from. Baseline as planned was presented for all participants/safety analysis set, skin cohort/analysis set and muscle cohort/analysis set.
Groups:
- PF-06823859 600mg: All Participants: Participants with DM received PF-06823859 600 mg IV once every 4 weeks. The treatment duration was up to 48 weeks (treatment period was up through and including Week 52). There was a follow-up period of 16 weeks post treatment period, however participants were assessed for safety from Day 1 of treatment up to end of study (Week 68).
Arm/Group | PF-06823859 600mg: All Participants
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Here, Number analyzed refers to number of participants analyzed per row.
  Years
    All Participants | 49.79 (12.73)
    Skin Cohort: number analyzed (Participants) | 9
    Skin Cohort | 51.78 (10.32)
    Muscle Cohort: number analyzed (Participants) | 15
    Muscle Cohort | 48.60 (14.19)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Here, Number analyzed refers to number of participants analyzed per row.
  Participants
    All Participants: Female | 20
    All Participants: Male | 4
    Skin Cohort: number analyzed (Participants) | 9
    Skin Cohort: Female | 9
    Skin Cohort: Male | 0
    Muscle Cohort: number analyzed (Participants) | 15
    Muscle Cohort: Female | 11
    Muscle Cohort: Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Here, Number analyzed refers to number of participants analyzed per row.
  Participants
    All Participants: Hispanic or Latino | 5
    All Participants: Not Hispanic or Latino | 19
    All Participants: Unknown or Not Reported | 0
    Skin Cohort: number analyzed (Participants) | 9
    Skin Cohort: Hispanic or Latino | 1
    Skin Cohort: Not Hispanic or Latino | 8
    Skin Cohort: Unknown or Not Reported | 0
    Muscle Cohort: number analyzed (Participants) | 15
    Muscle Cohort: Hispanic or Latino | 4
    Muscle Cohort: Not Hispanic or Latino | 11
    Muscle Cohort: Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Here, Number analyzed refers to number of participants analyzed per row.
  Participants
    All Participants: American Indian or Alaska Native | 0
    All Participants: Asian | 0
    All Participants: Native Hawaiian or Other Pacific Islander | 0
    All Participants: Black or African American | 0
    All Participants: White | 24
    All Participants: More than one race | 0
    All Participants: Unknown or Not Reported | 0
    Skin Cohort: number analyzed (Participants) | 9
    Skin Cohort: American Indian or Alaska Native | 0
    Skin Cohort: Asian | 0
    Skin Cohort: Native Hawaiian or Other Pacific Islander | 0
    Skin Cohort: Black or African American | 0
    Skin Cohort: White | 9
    Skin Cohort: More than one race | 0
    Skin Cohort: Unknown or Not Reported | 0
    Muscle Cohort: number analyzed (Participants) | 15
    Muscle Cohort: American Indian or Alaska Native | 0
    Muscle Cohort: Asian | 0
    Muscle Cohort: Native Hawaiian or Other Pacific Islander | 0
    Muscle Cohort: Black or African American | 0
    Muscle Cohort: White | 15
    Muscle Cohort: More than one race | 0
    Muscle Cohort: Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An Adverse Event (AE) was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE was considered treatment emergent relative to a given treatment if the event occurred for the first time during the effective duration of treatment and was not seen prior to the start of treatment, or the event was seen prior to the start of treatment but increased in severity during treatment. AEs included both serious adverse events (SAEs) and all non-SAEs.
Time Frame: From Day 1 of dosing maximum up to Week 68
Population: Safety Analysis Set included all participants enrolled who took at least 1 dose of study intervention, regardless of which stage the participant entered from. In this outcome measure data was planned to be reported for skin cohort/analysis set, muscle cohort/analysis set and all participants/safety analysis set.
Measure: Count of Participants; unit: Participants
Groups:
- PF-06823859 600mg: Skin Cohort: Participants with skin predominant DM entering from amended stage 2 of study C0251002 [NCT03181893] received PF-06823859 600 mg IV once every 4 weeks. The treatment duration was up to 48 weeks (treatment period was up through and including Week 52). There was a follow-up period of 16 weeks post treatment period, however participants were assessed for safety from Day 1 of treatment up to end of study (Week 68).
- PF-06823859 600mg: Muscle Cohort: Participants with muscle predominant DM entering from stage 3 of study C0251002 [NCT03181893] received PF-06823859 600 mg IV once every 4 weeks. The treatment duration was up to 48 weeks (treatment period was up through and including Week 52). There was a follow-up period of 16 weeks post treatment period, however participants were assessed for safety from Day 1 of treatment up to end of study (Week 68).
Arm/Group | PF-06823859 600mg: Skin Cohort | PF-06823859 600mg: Muscle Cohort | PF-06823859 600mg: All Participants
Number analyzed (Participants) | 9 | 15 | 24
Participants | 7 | 13 | 20

2. Primary Outcome: Number of Participants With Laboratory Abnormalities
Description: Hematology laboratory parameters: hemoglobin (grams per deciliter [g/dL]); hematocrit (percentage [%]); lymphocytes (10^3 per (/) millimeter[mm]^3); lymphocytes/leukocytes (%); neutrophils (10^3/mm^3) less than (<)0.8*lower limit of normal (LLN), leukocytes (10^3/mm^3) <0.6*LLN, neutrophils (10^3/mm^3); basophils (10^3/mm^3); basophils/leukocytes (%); monocytes/leukocytes (%); activated partial thromboplastin time (seconds [sec]); prothrombin time (sec) more than (>)1.2*upper limit of normal (ULN). Clinical chemistry: potassium (milliequivalents per liter [mEq/L]); bicarbonate (mEq/L) <0.9*LLN, creatine kinase (units per liter [U/L]) >2.0*ULN, glucose (milligram per deciliter [mg/dl]); glucose-fasting (mg/dl) >1.5*ULN. Urinalysis: Urine glucose; ketones; urine protein; urine hemoglobin; nitrite; leukocyte esterase; hyaline casts (1/per leukocytosis promoting factor (more than or equal to [>=] 1, urine erythrocytes (scalar); urine leukocytes (scalar) >=20.
Time Frame: From Day 1 of dosing maximum up to Week 68
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06823859 600mg: Skin Cohort | PF-06823859 600mg: Muscle Cohort | PF-06823859 600mg: All Participants
Number analyzed (Participants) | 9 | 15 | 24
Participants | 8 | 14 | 22

3. Primary Outcome: Number of Participants According to Categorization of Changes in Vital Signs
Description: Vital signs included the following parameters: sitting diastolic blood pressure (millimetres of mercury [mmHg]) change >=20 mmHg increase; sitting systolic blood pressure (mmHg) change >=30 mmHg increase, sitting diastolic blood pressure (mmHg) change >=20 mmHg decrease and sitting systolic blood pressure (mmHg) change >=30 mmHg decrease.
Time Frame: From Day 1 of dosing maximum up to Week 68
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06823859 600mg: Skin Cohort | PF-06823859 600mg: Muscle Cohort | PF-06823859 600mg: All Participants
Number analyzed (Participants) | 9 | 15 | 24
Participants
  Increase: sitting diastolic blood pressure (mmHg) | 4 | 4 | 8
  Increase: sitting systolic blood pressure (mmHg) | 4 | 2 | 6
  Decrease: sitting diastolic blood pressure (mmHg) | 1 | 4 | 5
  Decrease: sitting systolic blood pressure (mmHg) | 1 | 3 | 4

4. Primary Outcome: Number of Participants According to Categorization of Electrocardiogram (ECG) Findings
Description: ECG parameters evaluated were: PR interval value >=300 milliseconds (msec); QRS duration value >=200 msec; QT interval value >=500 msec; corrected QT Interval using Fridericia's formula (QTCF) 450 less than or equal to (<=) value <480 msec, 480 <=value<500 msec and value>=500 msec.
Time Frame: From Day 1 of dosing maximum up to Week 68
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06823859 600mg: Skin Cohort | PF-06823859 600mg: Muscle Cohort | PF-06823859 600mg: All Participants
Number analyzed (Participants) | 9 | 15 | 24
Participants
  PR interval: value >=300 msec | 0 | 0 | 0
  QRS duration: value >=200 msec | 0 | 0 | 0
  QT interval: >=500 msec | 0 | 0 | 0
  QTCF: 450<=value<480 msec | 2 | 1 | 3
  QTCF: 480<=value<500 msec | 0 | 0 | 0
  QTCF: value>=500 msec | 0 | 0 | 0

5. Secondary Outcome: Change From Baseline in Cutaneous Dermatomyositis Disease Area and Severity Index (CDASI) Activity Score at Week 52
Description: CDASI is a validated DM-specific instrument designed to systematically quantify the extent of cutaneous disease. Disease involvement in 15 different anatomical locations was rated using three activity (erythema, scale, erosion/ulceration) and two damage (poikiloderma, calcinosis) measures. The presence and severity of Gottron's papules, periungual changes and alopecia were also captured. Total CDASI activity score was based on the physician's evaluation of three activities (erythema, scale, erosion/ulceration), presence and severity of Gottron's papules, periungual changes and alopecia. Total CDASI activity score ranged from 0 to 100, where higher scores indicated higher levels of disability.
Time Frame: Baseline (before dose 1), Week 52
Population: Safety Analysis Set included all participants enrolled who took at least 1 dose of study intervention, regardless of which stage the participant entered from. In this outcome measure data was planned to be reported for skin cohort/analysis set and muscle cohort/analysis set. Here, "Number of Participants Analyzed" signifies number evaluable for this outcome measure.
Measure: Least Squares Mean (90% Confidence Interval); unit: Units on a scale
Arm/Group | PF-06823859 600mg: Skin Cohort | PF-06823859 600mg: Muscle Cohort
Number analyzed (Participants) | 9 | 12
Units on a scale | -4.67 [-7.41 to -1.92] | -2.51 [-3.40 to -1.62]

6. Secondary Outcome: Change From Baseline in CDASI Activity Score at Weeks 12, 24, 36, and 48
Description: as for outcome 5
Time Frame: Baseline (before dose 1), Weeks 12, 24, 36 and 48
Population: Safety Analysis Set included all participants enrolled who took at least 1 dose of study intervention, regardless of which stage the participant entered from. In this outcome measure data was planned to be reported for skin cohort/analysis set and muscle cohort/analysis set. Here "Number Analyzed" signifies number of participants evaluable for specified rows.
Measure: Least Squares Mean (90% Confidence Interval); unit: Units on a scale
Arm/Group | PF-06823859 600mg: Skin Cohort | PF-06823859 600mg: Muscle Cohort
Number analyzed (Participants) | 9 | 15
Units on a scale
  Change at Week 12: number analyzed (Participants) | 8 | 15
  Change at Week 12 | -5.28 [-7.67 to -2.90] | -0.87 [-1.98 to 0.25]
  Change at Week 24 | -4.11 [-6.47 to -1.75] | -0.67 [-2.09 to 0.75]
  Change at Week 36: number analyzed (Participants) | 8 | 15
  Change at Week 36 | -4.51 [-7.90 to -1.11] | -1.40 [-2.40 to -0.40]
  Change at Week 48: number analyzed (Participants) | 9 | 12
  Change at Week 48 | -4.56 [-7.27 to -1.84] | -1.70 [-2.70 to -0.70]

7. Secondary Outcome: Absolute Values of CDASI Activity Score at Weeks 12, 24, 36, 48, and 52
Description: as for outcome 5
Time Frame: Weeks 12, 24, 36, 48 and 52
Population: Safety Analysis Set included all participants enrolled who took at least 1 dose of study intervention, regardless of which stage the participant entered from. In this outcome measure data was planned to be reported for skin cohort/analysis set and muscle cohort/analysis set. Here, "Number Analyzed" signifies number evaluable for specified rows.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | PF-06823859 600mg: Skin Cohort | PF-06823859 600mg: Muscle Cohort
Number analyzed (Participants) | 9 | 15
Units on a scale
  Week 12: number analyzed (Participants) | 8 | 15
  Week 12 | 4.4 (2.45) | 4.4 (3.44)
  Week 24 | 5.0 (3.71) | 4.6 (3.81)
  Week 36: number analyzed (Participants) | 8 | 15
  Week 36 | 5.5 (5.13) | 3.9 (3.27)
  Week 48: number analyzed (Participants) | 9 | 12
  Week 48 | 4.6 (4.45) | 3.1 (3.03)
  Week 52: number analyzed (Participants) | 9 | 12
  Week 52 | 4.4 (4.85) | 2.2 (2.52)

8. Secondary Outcome: Change From Baseline in CDASI Damage Score at Weeks 12, 24, 36, 48, and 52
Description: CDASI is a validated DM-specific instrument designed to systematically quantify the extent of cutaneous disease. Disease involvement in 15 different anatomical locations was rated using three activity (erythema, scale, erosion/ulceration) and two damage (poikiloderma, calcinosis) measures. The presence and severity of Gottron's papules, periungual changes and alopecia were also captured. Total CDASI damage score was based on the physician's evaluation of two damage (poikiloderma, calcinosis) measures, and presence and severity of Gottron's papules. Total CDASI damage score ranged from 0 to 32, where higher scores indicated higher level of skin damage.
Time Frame: Baseline (before dose on Day 1), Weeks 12, 24, 36, 48 and 52
Population: Safety Analysis Set included all participants enrolled who took at least 1 dose of study intervention, regardless of which stage the participant entered from. In this outcome measure data was planned to be reported for skin cohort/analysis set and muscle cohort/analysis set. Here "Number Analyzed" signifies number evaluable for specified rows.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | PF-06823859 600mg: Skin Cohort | PF-06823859 600mg: Muscle Cohort
Number analyzed (Participants) | 9 | 15
Units on a scale
  Change at Week 12: number analyzed (Participants) | 8 | 15
  Change at Week 12 | -2.4 (2.77) | -0.8 (1.15)
  Change at Week 24 | -1.8 (2.33) | -0.5 (1.19)
  Change at Week 36: number analyzed (Participants) | 8 | 15
  Change at Week 36 | -2.3 (2.25) | -0.5 (1.06)
  Change at Week 48 | -2.0 (2.00) | -0.9 (1.24)
  Change at Week 52 | -2.1 (2.09) | -0.9 (1.08)

9. Secondary Outcome: Absolute Values of CDASI Damage Score at Weeks 12, 24, 36, 48, and 52
Description: as for outcome 8
Time Frame: Weeks 12, 24, 36, 48 and 52
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | PF-06823859 600mg: Skin Cohort | PF-06823859 600mg: Muscle Cohort
Number analyzed (Participants) | 9 | 15
Units on a scale
  Week 12: number analyzed (Participants) | 8 | 15
  Week 12 | 0.9 (1.25) | 1.6 (3.07)
  Week 24 | 1.9 (2.26) | 1.9 (3.41)
  Week 36: number analyzed (Participants) | 8 | 15
  Week 36 | 1.4 (2.33) | 1.9 (3.43)
  Week 48: number analyzed (Participants) | 9 | 12
  Week 48 | 1.7 (2.12) | 1.3 (2.83)
  Week 52: number analyzed (Participants) | 9 | 12
  Week 52 | 1.6 (1.59) | 1.3 (3.19)

10. Secondary Outcome: Total Improvement Score (TIS) at Weeks 12, 24, 36, 48 and 52: Muscle Cohort
Description: There are 6 core set measure that comprised of TIS: 1) Physician Global Assessment Score [PhGA] (from Myositis Disease Activity Assessment Tool [MDAAT], 0-100 mm or 0-10 centimeter (cm) on visual analogue scale [VAS], higher scores= worse health status); 2) Patient Global Assessment Score [PtGA] (0-100 mm or 0-10 cm on VAS, higher scores= worse status); 3) Manual Muscle Testing-8 (MMT-8) designated muscle groups (0-80, lower scores= higher level of disability); 4) Health Assessment Questionnaire Disability Index [HAQ-DI] (0-3, higher scores= worse status); 5) Global Extramuscular Disease Activity (from MDAAT, 0-10 cm on a VAS, higher scores= higher level of disability); 6) Participant's most elevated muscle enzymes. TIS was sum of all 6 improvement scores associated with the change in each core set measure. TIS ranged from 0 to 100; where TIS>=20 shows minimal improvement, TIS >=40 shows moderate improvement and TIS >= 60 shows major improvement.
Time Frame: Weeks 12, 24, 36, 48 and 52
Population: Safety Analysis Set included all participants enrolled who took at least 1 dose of study intervention, regardless of which stage the participant entered from. In this outcome measure data was planned to be reported for muscle cohort/analysis set. Here "Number Analyzed" signifies number evaluable for specified rows.
Measure: Least Squares Mean (90% Confidence Interval); unit: Units on a scale
Arm/Group | PF-06823859 600mg: Muscle Cohort
Number analyzed (Participants) | 15
Units on a scale
  Week 12: number analyzed (Participants) | 14
  Week 12 | 15.03 [8.36 to 21.70]
  Week 24 | 15.67 [8.96 to 22.37]
  Week 36 | 18.17 [10.84 to 25.49]
  Week 48: number analyzed (Participants) | 12
  Week 48 | 19.61 [10.58 to 28.63]
  Week 52: number analyzed (Participants) | 12
  Week 52 | 23.66 [14.05 to 33.28]

11. Secondary Outcome: Change From Baseline in Physician Global Assessment (PhGA) Score at Week 12, 24, 36, 48 and 52: Muscle Cohort
Description: PhGA: Investigator was asked to evaluate the participant's overall disease activity on a VAS of 0 cm (very good) to 10 cm (very poor), higher scores indicated worse health status.
Time Frame: Baseline (before dose on day 1), Weeks 12, 24, 36, 48 and 52
Population: as for outcome 10
Measure: Least Squares Mean (90% Confidence Interval); unit: centimeter
Arm/Group | PF-06823859 600mg: Muscle Cohort
Number analyzed (Participants) | 15
centimeter
  Change at Week 12: number analyzed (Participants) | 14
  Change at Week 12 | 0.17 [-0.54 to 0.87]
  Change at Week 24 | 0.29 [-0.39 to 0.98]
  Change at Week 36 | -0.18 [-0.59 to 0.23]
  Change at Week 48: number analyzed (Participants) | 12
  Change at Week 48 | -0.48 [-0.85 to -0.10]
  Change at Week 52: number analyzed (Participants) | 12
  Change at Week 52 | -0.60 [-0.97 to -0.23]

12. Secondary Outcome: Change From Baseline in Patient Global Assessment (PtGA) Score at Weeks 12, 24, 36, 48 and 52: Muscle Cohort
Description: PtGA was the assessment of the severity of disease by the participant/participant's guardian, using a VAS from 0 mm (no evidence of disease activity) to 100 mm (extremely active or severe disease activity). Higher score indicated worse status.
Time Frame: Baseline (before dose on day 1), Weeks 12, 24, 36, 48 and 52
Population: as for outcome 10
Measure: Least Squares Mean (90% Confidence Interval); unit: millimeter
Arm/Group | PF-06823859 600mg: Muscle Cohort
Number analyzed (Participants) | 15
millimeter
  Change at Week 12 | 3.70 [-6.55 to 13.95]
  Change at Week 24 | -9.63 [-18.18 to -1.08]
  Change at Week 36 | -9.10 [-16.47 to -1.73]
  Change at Week 48: number analyzed (Participants) | 12
  Change at Week 48 | -8.36 [-14.74 to -1.97]
  Change at Week 52: number analyzed (Participants) | 12
  Change at Week 52 | -6.28 [-16.79 to 4.22]

13. Secondary Outcome: Change From Baseline in Manual Muscle Testing-8 Designated Muscle Groups (MMT-8) Score at Weeks 12, 24, 36, 48 and 52: Muscle Cohort
Description: MMT-8 is a tool that assesses muscle strength using manual muscle testing. Eight designated muscles are tested unilaterally with a total potential summed score of 0-80. Lower scores indicated a higher level of disability.
Time Frame: Baseline (before dose on day 1), Weeks 12, 24, 36, 48 and 52
Population: as for outcome 10
Measure: Least Squares Mean (90% Confidence Interval); unit: Units on a scale
Arm/Group | PF-06823859 600mg: Muscle Cohort
Number analyzed (Participants) | 15
Units on a scale
  Change at Week 12: number analyzed (Participants) | 14
  Change at Week 12 | -0.06 [-5.93 to 5.82]
  Change at Week 24 | 1.85 [-3.11 to 6.81]
  Change at Week 36 | 4.92 [0.61 to 9.22]
  Change at Week 48: number analyzed (Participants) | 12
  Change at Week 48 | 8.00 [5.69 to 10.30]
  Change at Week 52: number analyzed (Participants) | 12
  Change at Week 52 | 9.84 [7.38 to 12.31]

14. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire and Disease Index (HAQ-DI) Score at Weeks 12, 24, 36, 48 and 52: Muscle Cohort
Description: HAQ-DI consisted of eight sections (including dressing & grooming, arising, eating, walking, hygiene, grip, reach, and activities). Each section had multiple questions that the participant used to rank their functionality and ranged from 0 to 3 where 0 = without any difficulty and 3 = unable to do. For each participant, the average ranking was calculated for each of the eight sections. HAQ-DI had a score range of 0 to 3, where higher score reflected worse status.
Time Frame: Baseline (before dose on day 1), Weeks 12, 24, 36, 48 and 52
Population: as for outcome 10
Measure: Least Squares Mean (90% Confidence Interval); unit: Units on a scale
Arm/Group | PF-06823859 600mg: Muscle Cohort
Number analyzed (Participants) | 15
Units on a scale
  Change at Week 12 | 0.00 [-0.13 to 0.13]
  Change at Week 24 | -0.10 [-0.21 to 0.01]
  Change at Week 36 | -0.07 [-0.23 to 0.08]
  Change at Week 48: number analyzed (Participants) | 12
  Change at Week 48 | -0.12 [-0.24 to 0.00]
  Change at Week 52: number analyzed (Participants) | 12
  Change at Week 52 | -0.18 [-0.32 to -0.04]

15. Secondary Outcome: Change From Baseline in Creatine Kinase at Weeks 12, 24, 36, 48 and 52: Muscle Cohort
Description: Creatine kinase is a muscle enzyme measured in units per liter (U/L).
Time Frame: Baseline (before dose on day 1), Weeks 12, 24, 36, 48 and 52
Population: as for outcome 10
Measure: Least Squares Mean (90% Confidence Interval); unit: Units per liter
Arm/Group | PF-06823859 600mg: Muscle Cohort
Number analyzed (Participants) | 15
Units per liter
  Change at Week 12 | -98.93 [-163.76 to -34.11]
  Change at Week 24 | -58.53 [-127.24 to 10.17]
  Change at Week 36: number analyzed (Participants) | 14
  Change at Week 36 | -97.62 [-150.82 to -44.42]
  Change at Week 48: number analyzed (Participants) | 12
  Change at Week 48 | -72.04 [-161.48 to 17.39]
  Change at Week 52: number analyzed (Participants) | 12
  Change at Week 52 | -94.04 [-147.13 to -40.95]

16. Secondary Outcome: Change From Baseline in Extramuscular Global Assessment From the Myositis Disease Activity Assessment Tool (MDAAT) Score at Weeks 12, 24, 36, 48 and 52: Muscle Cohort
Description: MDAAT tool measures the degree of disease activity of extramuscular organ systems and muscle on a VAS of 0 to 10 cm, higher scores indicated higher level of disability.
Time Frame: Baseline (before dose on day 1), Weeks 12, 24, 36, 48 and 52
Population: as for outcome 10
Measure: Least Squares Mean (90% Confidence Interval); unit: centimeter
Arm/Group | PF-06823859 600mg: Muscle Cohort
Number analyzed (Participants) | 15
centimeter
  Change at Week 12: number analyzed (Participants) | 14
  Change at Week 12 | 0.05 [-0.40 to 0.50]
  Change at Week 24 | 0.23 [-0.23 to 0.68]
  Change at Week 36 | 0.01 [-0.51 to 0.53]
  Change at Week 48: number analyzed (Participants) | 12
  Change at Week 48 | -0.16 [-0.91 to 0.59]
  Change at Week 52: number analyzed (Participants) | 12
  Change at Week 52 | -0.56 [-1.07 to -0.06]

ADVERSE EVENTS:
Time Frame: From Day 1 of dosing maximum up to Week 68
Description: Same event may appear as both non-SAE and SAE. What is presented are distinct events. An event may be categorized as serious in 1 participant and non-serious in other participant, or a participant may have experienced both SAE and non-SAE. Safety analysis set included all participants enrolled who had taken at least 1 dose of study intervention. This included all such participants regardless of which parent study or stage the participant entered from.
Arm/Group | PF-06823859 600mg: Skin Cohort | PF-06823859 600mg: Muscle Cohort | PF-06823859 600mg: All Participants
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/15 | 0/24
Serious Adverse Events (participants affected / at risk) | 1/9 | 2/15 | 3/24
Other Adverse Events (participants affected / at risk) | 7/9 | 13/15 | 20/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-06823859 600mg: Skin Cohort (N=9) | PF-06823859 600mg: Muscle Cohort (N=15) | PF-06823859 600mg: All Participants (N=24)
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-06823859 600mg: Skin Cohort (N=9) | PF-06823859 600mg: Muscle Cohort (N=15) | PF-06823859 600mg: All Participants (N=24)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 2
Palpitations (Cardiac disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1
Faeces discoloured (Gastrointestinal disorders) | 0 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Calcinosis (General disorders) | 0 | 1 | 1
Chest discomfort (General disorders) | 0 | 1 | 1
Infusion site extravasation (General disorders) | 1 | 0 | 1
Infusion site rash (General disorders) | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 1 | 1
Bronchitis (Infections and infestations) | 1 | 1 | 2
COVID-19 (Infections and infestations) | 3 | 3 | 6
Cystitis (Infections and infestations) | 1 | 0 | 1
Fungal infection (Infections and infestations) | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 1
Herpes zoster (Infections and infestations) | 0 | 1 | 1
Influenza (Infections and infestations) | 0 | 1 | 1
Laryngitis (Infections and infestations) | 1 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 1
Respiratory tract infection viral (Infections and infestations) | 1 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 1 | 2
Tooth infection (Infections and infestations) | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 2 | 3
Vulvovaginal candidiasis (Infections and infestations) | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1
Sunburn (Injury, poisoning and procedural complications) | 0 | 1 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Blood potassium decreased (Investigations) | 1 | 0 | 1
Blood pressure increased (Investigations) | 1 | 0 | 1
Crystal urine present (Investigations) | 0 | 1 | 1
Weight increased (Investigations) | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 2 | 2
Mental impairment (Nervous system disorders) | 0 | 1 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1 | 1
Renal colic (Renal and urinary disorders) | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Cutaneous calcification (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Nail pigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Hypotension (Vascular disorders) | 1 | 0 | 1
Lymphoedema (Vascular disorders) | 1 | 0 | 1
Peripheral venous disease (Vascular disorders) | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-09-03): https://cdn.clinicaltrials.gov/large-docs/00/NCT05192200/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-30): https://cdn.clinicaltrials.gov/large-docs/00/NCT05192200/SAP_001.pdf